CLINICAL TRIAL: NCT02877875
Title: Student Outcomes of Integrative Mental Health Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, John Weisz, Professor and Principal Investigator, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R305A140253
Record Dates: First submitted 2015-01-06; First posted 2016-08-24 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Anxiety; Depression; Trauma; Behavior Problems
Keywords: anxiety; depression; trauma; behavior problems; evidence-based treatments; manualized treatments; cognitive-behavioral therapy; youth; mental health
MeSH Terms: conditions — Anxiety Disorders; Depression; Wounds and Injuries; Mental Disorders; Psychological Well-Being | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Child STEPS (Experimental): Child STEPs includes (1) a treatment protocol, Modular Approach to Therapy for Children with Anxiety, Depression, Trauma or Conduct Problems (MATCH-ADTC;Chorpita & Weisz, 2009), and (2) a youth monitoring and feedback system (MFS).
  Interventions: Behavioral: Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, and Conduct Problems; Other: Monitoring and Feedback System
- Usual Care (Active Comparator): Treatment in the UC condition will use the procedures therapists and their supervisors consider appropriate and believe to be effective, and researchers will not influence their work.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, and Conduct Problems — MATCH-ADTC (Chorpita & Weisz, 2009) is designed for children aged 6-15. Unlike most evidence-based treatments (EBTs), which focus on single disorder categories (e.g., anxiety only), MATCH is designed for multiple disorders and problems encompassing anxiety, depression, post-traumatic stress, and disruptive conduct, including the conduct problems associated with Attention-deficit/hyperactivity disorder (ADHD). MATCH is composed of 33 modules-i.e., specific treatment procedures derived from decades of research on EBTs. The various modules can be organized and sequenced flexibly to tailor treatment to each child's characteristics and needs.
  Other Names: MATCH; MATCH - ADTC
  Arms: Child STEPS
Other: Monitoring and Feedback System — For each child, the web-based MFS system provides weekly monitoring of the MATCH modules used and the child's treatment response, in two forms (a) changes on the Behavior and Feelings Survey and (b) changes in severity of the top treatment concerns identified by youths and caregivers. At the end of treatment, the MFS provides a complete record of modules used, and child treatment response, across all the weeks of treatment.
  Other Names: MFS
  Arms: Child STEPS
Behavioral: Treatment as usual — Treatment in the UC condition will use the procedures therapists (e.g., school counselors) and their supervisors consider appropriate and believe to be effective.
  Other Names: Usual Care; UC
  Arms: Usual Care

SUMMARY:
The study will compare the impact of Child STEPs (see Weisz et al., 2012) versus usual school-based therapy on students' mental health and school-related outcomes, and test whether changes in school outcomes are mediated by changes in student mental health.

DETAILED DESCRIPTION:
This project will implement and evaluate the Child STEPs (see Weisz et al., 2012) treatment approach through a randomized controlled trial (RCT) at 27 K-8 public schools. The STEPs model has two components: (1) a modular protocol that combines 33 modules-i.e., descriptions of common elements within evidence-based therapies for anxiety, depression, post-traumatic stress, and conduct problems; and (2) a web-based system for monitoring student responses to treatment and providing weekly feedback to therapists, to guide their selection and sequencing of the STEPs modules. The project will include an evaluation of the effectiveness of STEPS compared to "treatment as usual" (known as Usual Care or UC) on students' mental health and school-related outcomes, and an analysis of whether changes in school outcomes are mediated by changes in student mental health.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in grades 2-7
2. Have a primary clinical problem in the areas of anxiety, depression, conduct, or posttraumatic stress
3. Clinically elevated problem levels on the Internalizing, Externalizing, Anxious-Depressed, Withdrawn-Depressed, Aggressive Behavior, or Rule-Breaking Behavior scales of the Child Behavior Checklist or Youth Self-Report or on the UCLA Post-traumatic Stress Disorder Reaction Index

Exclusion Criteria:

1. Mental retardation
2. Pervasive developmental disorder
3. Eating disorders
4. Children for whom attention problems or hyperactivity are the primary referral concern
5. Active psychosis and/or a suicide attempt in the previous year

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 143 (Actual)
Dates: Start 2015-01; Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Change in internalizing and externalizing problems per self- and caregiver-report. | Change over time from Baseline (Day 1) through study completion (up to 66 weeks)
  The Behavior and Feelings Survey-Youth and Caregiver Report (BFS-Youth and Caregiver) is a no-cost, 12-item, youth- and caregiver-report measure of internalizing and externalizing problems. The BFS-Youth and Caregiver showed robust factor structure, internal consistency, test-retest reliability, and slopes of change indicating efficacy in monitoring treatment progress during psychotherapy in four samples of youths aged 7-15 years. The BFS-Youth and Caregiver is administered weekly.
Change in internalizing and externalizing problems per teacher-report. | Change over time from Baseline (Day 1) through post-treatment (up to 34 weeks)
  The Behavior and Feelings Survey-Teacher Report (BFS-Teacher) is a no-cost, 12-item, teacher-report measure of internalizing and externalizing problems. The BFS-Teacher showed robust factor structure, internal consistency, test-retest reliability, and slopes of change indicating efficacy in monitoring treatment progress during psychotherapy in four samples of youths aged 7-15 years. The BFS-Teacher is administered monthly.
Change in top problems per youth- and caregiver-report. | Change over time from Baseline (Day 1) through study completion (up to 66 weeks)
  The Top Problems Assessment-Youth and Caregiver Report (TPA- Youth and Caregiver) is a brief idiographic instrument designed to help identify and monitor youth problems that are especially important from the perspectives of the youth and caregiver. The TPA- Youth and Caregiver were shown to complement standardized measures and offer incremental utility, with evidence of test- retest reliability, convergent and discriminant validity, and sensitivity to change during treatment. The TPA-Youth and Caregiver is administered weekly.
Change in top problems per teacher-report. | Change over time from Baseline (Day 1) through Post-treatment (up to 34 weeks)
  The Top Problems Assessment-Teacher Report (TPA-Teacher) is a brief idiographic instrument designed to help identify and monitor youth problems that are especially important from the perspectives of the youth's teacher. The TPA-Teacher has not yet been examined psychometrically. The TPA-Youth and Caregiver is administered monthly.
Academic outcomes, assessed via school grades and standardized test performance | Yearly, assessed up to 52 weeks
  Academic outcomes as obtained through class grades and standardized school testing.
Change in school engagement per self- and caregiver-report. | Change over time from Baseline (Day 1) through study completion (up to 66 weeks)
  The National Survey of American Families (NSAF-Youth and Caregiver) School Engagement Scale is a youth- and caregiver-reported is a measure of behavioral, emotional, and cognitive engagement in school. Respondents rate youth on a four-point scale on items assessing whether the youth cares about doing well in school, only works on schoolwork when forced to, does just enough schoolwork to get by, and always does their homework
Change in school engagement per teacher-report. | Change over time from Baseline (Day 1) through Post-treatment (up to 34 weeks)
  The National Survey of American Families (NSAF-Teacher) School Engagement Scale is a measure of behavioral, emotional, and cognitive engagement in school. Respondents rate youth on a four-point scale on items assessing whether the youth cares about doing well in school, only works on schoolwork when forced to, does just enough schoolwork to get by, and always does their homework. NSAF-Teacher is administered monthly.

SECONDARY OUTCOMES:
Youth Self-Report (YSR) | Change over time from Baseline (Day 1) through study completion (up to 66 weeks)
  Self-report measure of child behavioral and emotional problems. Each item is rated 0 (Not True), 1 (Somewhat or Sometimes True), or 2 (Very True or Often True). Measure generates a total problems scale, broadband Internalizing and Externalizing syndrome scales, and eight narrowband syndrome scales (e.g., Aggressive Behavior). The YSR is supported by extensive psychometric evidence. Youth complete the YSR at baseline, post-treatment, and 6 month follow-up.
Child Behavior Checklist (CBCL) | Change over time from Baseline (Day 1) through study completion (up to 66 weeks)
  Caregiver-report measure of child behavioral and emotional problems. Each item is rated 0 (Not True), 1 (Somewhat or Sometimes True), or 2 (Very True or Often True). Measure generates a total problems scale, broadband Internalizing and Externalizing syndrome scales, and eight narrowband syndrome scales (e.g., Aggressive Behavior). The CBCL is supported by extensive psychometric evidence. Caregivers complete the CBCL at baseline, post-treatment, and 6 month follow-up.
Teacher Report Form (TRF) | Change over time from Baseline (Day 1) to Post-treatment (up to 34 weeks)
  Teacher-report measure of child behavioral and emotional problems. Each item is rated 0 (Not True), 1 (Somewhat or Sometimes True), or 2 (Very True or Often True). Measure generates a total problems scale, broadband Internalizing and Externalizing syndrome scales, and eight narrowband syndrome scales (e.g., Aggressive Behavior). The TRF is supported by extensive psychometric evidence.
University of California at Los Angeles (UCLA) Post-traumatic Stress Disorder Reaction Index | Change over time from Baseline (Day 1) through study completion (up to 66 weeks)
  This 38-item measure is widely-used to assess child post-traumatic stress symptoms. Part I is a brief lifetime trauma screen. If the participant identifies significant trauma, Part II assesses Diagnostic and Statistical Manual-IV (DSM-IV) PTSD symptoms related to the trauma. Part III assesses frequency of post-traumatic stress symptoms during the past month. The UCLA Post-traumatic Stress Disorder Reaction Index is administered separately to youth and their caregivers at baseline, post-treatment, and 6 month follow-up.
Services Assessment for Children and Adolescents (SACA) | Baseline (Day 1) through study completion (up to 66 weeks)
  To assess whether treatment reduced the need for other services, a modified version of the Services Assessment for Children and Adolescents (SACA), a standardized parent-report interview assessing use of multiple mental health services (e.g., medication for a behavioral or emotional problem, inpatient psychiatric hospitalization) will be administered. At pre-treatment, the reporting time frame will be the previous 6 months, to establish a baseline for each student; at post-treatment, the time frame will be the period when treatment was received; at follow-up, the time frame will be the 6 months since treatment ended.
Medication Questionnaire adapted from the Services for Children and Adolescents-Parent Interview (SCA-PI) | Baseline (Day 1) through study completion (up to 66 weeks)
  To assess whether medication influenced students' intervention response, we ask caregivers a series of questions to assess medications, dosage, and reasons for the medications--adapted from the SCA-PI (a standardized parent-report interview). The SCA-PI has particular strength in medication assessment, including start dates, end dates, and dosage. The medication questionnaire is administered at baseline, post-treatment, and at 6-month follow-up.
Therapeutic Alliance Scale (TASC) | Post-treatment, assessed up to 42 weeks after baseline
  Youth and caregivers will be given the TASC, to assess the quality of the youth's working alliance with the therapist.This 7-item scale comes in both a youth-report form and a parent-report form (parents reporting on their youth's relationship with the therapist).
Caregiver Satisfaction Questionnaire | Post-treatment, assessed up to 42 weeks after baseline
  Caregivers complete the Caregiver Satisfaction Questionnaire at post-treatment, assessed up to 40 weeks after baseline. The Caregiver Satisfaction Questionnaire is 8 questions (e.g., "How would you rate the quality of the counseling services that were provided?").
Youth Satisfaction Questionnaire | Post-treatment, assessed up to 42 weeks after baseline
  The Youth Satisfaction Questionnaire consists of 8 questions (e.g., "Overall, how happy are you with the help you got?") assessing the youth's satisfaction with mental health services.
Therapist Satisfaction Inventory (TSI) | Post-treatment, assessed up to 42 weeks after baseline
  Therapists complete the TSI at the completion of treatment. The TSI is a 16-item measure that assesses whether therapists liked the treatment approach they used, whether the approach made them feel effective, whether they believe it allowed them to individualize treatment to fit the needs of the client, and whether it seems appropriate for the kinds of children they most often see.
Emotion Regulation Checklist (ERC) | Change over time from Baseline (Day 1) through study completion (up to 66 weeks)
  The ERC is a 24-item questionnaire using a 4-point Likert scale that assesses the caregiver's perceptions of their children's ability to manage emotion. This measure yields two empirically derived scales: (a) Emotion Regulation that assesses situationally appropriate affective displays and emotional self-awareness, and (b) Lability/Negativity, which measures mood lability and culturally inappropriate affective displays. Internal consistency has been established for this measure as well as support for its construct validity. Caregivers complete the ERC at baseline, post-treatment, and 6-month follow-up.
Brief Symptom Inventory (BSI) | Baseline (Day 1)
  Caregivers complete this 53-item, self-report measure of adult symptomatology at baseline. This measure generates scores on nine dimensions (e.g., Depression, Anxiety, Hostility) and a General Severity Index (GSI).
The Children's Emotion Management Scale (CEMS) | Change over time from Baseline (Day 1) through study completion (up to 66 weeks)
  The CEMS assesses children's self-report of sadness, anger, and worry regulation. Children indicate the frequency with which they engage in a variety of emotion management strategies using a Likert scale of 1 (hardly ever), 2 (sometimes), or 3 (often). Three subscales have been identified for each emotion: (a) Inhibition (four items),(b) Dysregulated Expression (three items), and (c) Emotion Regulation Coping (five items for sadness scale and four items for anger scale). Examination of the reliability of the CEMS anger and sadness scales indicate coefficient alphas that range from .62 to .77 and test-retest reliability ranging from .61 to .80 for the individual subscales. Children complete the CEMS at baseline, post-treatment, and 6 month follow-up.
The Children's Response Style Questionnaire (CRSQ) | Change over time from Baseline (Day 1) through study completion (up to 66 weeks)
  The CRSQ is modeled after Nolen-Hoeksema's Response Styles Questionnaire and consists of 25 items, each of which describes a particular response to symptoms of depression. The items are grouped into three scales: (1) Ruminative Response subscale (CRSQ-Rumination); (2) Distracting Response subscale (CRSQ-Distraction); and (3) Problem-Solving subscale (CRSQ-Problem solving). For each item, youth are asked to indicate how often they respond in this way when they are feeling sad (almost never = 0,sometimes = 1, often = 2, or almost always = 3). Scores range from 0 to 39 on the Ruminative Response subscale, from 0 to 21 on the Distracting Response subscale, and from 0 to 15 on the Problem Solving subscale. Higher scores on each subscale indicate a greater tendency to engage in that particular response style.Children complete the CRSQ at baseline, post-treatment, and at 6 month follow-up.
Perceived Control Scale for Children (PCSC) | Change over time from Baseline (Day 1) through study completion (up to 66 weeks)
  The PCSC assesses perceived ability to exert primary control -that is, to influence or alter objective events or conditions through one's own effort. Youth rate agreement with statements about their ability to exert primary control, with half the items worded in a positive direction (e.g., "I can do well on tests if I study hard.") and half in a negative direction (e.g., "I cannot get other kids to like me no matter how hard I try."). Responses can range from "very true" to "very false." This scale has shown acceptable internal consistency (α=0.88) and six-month test-retest reliability (r=0.57) as well as a strong inverse relation to depressive symptoms (r=0.58 with Children's Depression Inventory scores).
Secondary Control Scale for Children (SCSC) | Change over time from Baseline (Day 1) through study completion (up to 66 weeks)
  This 20-item scale was designed to assess perceived ability to exert secondary control-that is, to influence the personal psychological impact of objective conditions on oneself, by adjusting oneself to fit those conditions. The item content reflects response patterns associated with secondary control in the two-process model, for example, finding a silver lining, adjusting cognition, avoiding rumination, and generic secondary control. To discourage response sets, half the items are worded in a positive direction and half in a negative direction. Respondents rate their agreement with each item (on a 4-point scale, from "very false" to "very true").
Reduced Aggression and Victimization Scales (RAVS) | Change over time from Baseline (Day 1) through study completion (up to 66 weeks)
  The RAVS measures the frequency of reporting aggressive behaviors or of being victimized during the previous week prior to the survey. The scales are composed of six items each. Each point represents one instance of aggression or victimization reported by the child. The RAVS is administered at baseline, post-treatment, and 6 month follow-up.
Implicit Theories of Thoughts, Emotions, and Behaviors Scale (ITEB-Q) | Change over time from Baseline (Day 1) through study completion (up to 66 weeks)
  This study includes a new scale adapted from Dweck's work on implicit theories for intelligence to measure implicit theories regarding thoughts, emotions, and behaviors. The ITEB-Q contains twelve items; four items each address implicit theories regarding thoughts, feelings, and behavior. Items on each subscale present extreme incremental theory beliefs (e.g., "When I try, I can control how I feel," "When I feel bad, I can make myself feel better"). Responses are measured using a four-point scale ranging from 1 ("Very False") to 4 ("Very True"). The higher participants' summed scores on the full ITEB-Q, the less they believe thoughts, emotions, and behavior are fixed entities.
Children's Alexithymia Scale (CAS) | Change over time from Baseline (Day 1) through study completion (up to 66 weeks)
  The Children's Alexithymia Scale is based on the original Toronto Alexithymia Scale 20 that assesses alexithymia in adults.The Alexithymia Questionnaire for Children consists of 20 items that represent the three factors: Difficulty identifying feelings, Difficulty describing feelings and Externally oriented thinking. The item response format is: strongly disagree to strongly agree.
Evidence-Based Practice Attitudes Scale (EBPAS) | Change over time from Baseline (Day 1) to Post-treatment (up to 42 weeks)
  The EBPAS consists of 15 items measured on a 5-point scale ranging from 0 (Not at all) to 4 (To a very great extent). The EBPAS is comprised of four subscales (Appeal, Requirements, Openness, and Divergence) and a total scale score, which represents respondents' global attitude toward adoption of EBPs. Cronbach's alpha reliability for the EBPAS is good (alpha = 0.77), with subscale alphas ranging from 0.59 to 0.90.
Academic Competence Evaluation Scales | Change over time from Baseline (Day 1) to Post-treatment (up to 34 weeks)
  School functioning in the classroom will be assessed via the Academic Competence Evaluation Scales (ACES) is a 60-item, teacher-reported scale which assesses youth Academic Skills (including Reading/Language Arts, Mathematics, and Critical Thinking) and Academic Enablers (including Interpersonal Skills, Engagement, Motivation, and Study Skills). The ACES has demonstrated internal consistency and test-retest reliability.
The School Engagement Measure-MacArthur Network | Change over time from Baseline (Day 1) through study completion (up to 66 weeks)
  The School Engagement Measure-MacArthur Network is a youth-self report measure of three components of youth engagement that have been supported in factor analysis; these are: Behavioral, Emotional and Cognitive. The Cognitive subscale has not fared so well psychometrically, so only the two psychometrically stronger subscales: Behavioral and Emotional Engagement, will be administered to youth. Youth complete this measure at baseline, post-treatment, and 6 month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: John R. Weisz, Principal Investigator — Harvard University
Locations (1):
- Harvard University, Cambridge, Massachusetts, United States

REFERENCES:
- [Background] Weisz JR, Chorpita BF, Palinkas LA, Schoenwald SK, Miranda J, Bearman SK, Daleiden EL, Ugueto AM, Ho A, Martin J, Gray J, Alleyne A, Langer DA, Southam-Gerow MA, Gibbons RD; Research Network on Youth Mental Health. Testing standard and modular designs for psychotherapy treating depression, anxiety, and conduct problems in youth: a randomized effectiveness trial. Arch Gen Psychiatry. 2012 Mar;69(3):274-82. doi: 10.1001/archgenpsychiatry.2011.147. Epub 2011 Nov 7. PMID 22065252
- [Background] Weisz JR, Chorpita BF, Frye A, Ng MY, Lau N, Bearman SK, Ugueto AM, Langer DA, Hoagwood KE; Research Network on Youth Mental Health. Youth Top Problems: using idiographic, consumer-guided assessment to identify treatment needs and to track change during psychotherapy. J Consult Clin Psychol. 2011 Jun;79(3):369-80. doi: 10.1037/a0023307. PMID 21500888
- [Background] Goodman A, Lamping DL, Ploubidis GB. When to use broader internalising and externalising subscales instead of the hypothesised five subscales on the Strengths and Difficulties Questionnaire (SDQ): data from British parents, teachers and children. J Abnorm Child Psychol. 2010 Nov;38(8):1179-91. doi: 10.1007/s10802-010-9434-x. PMID 20623175
- [Background] Addis ME, Krasnow AD. A national survey of practicing psychologists' attitudes toward psychotherapy treatment manuals. J Consult Clin Psychol. 2000 Apr;68(2):331-9. doi: 10.1037//0022-006x.68.2.331. PMID 10780134
- [Background] Shields A, Cicchetti D. Emotion regulation among school-age children: the development and validation of a new criterion Q-sort scale. Dev Psychol. 1997 Nov;33(6):906-16. doi: 10.1037//0012-1649.33.6.906. PMID 9383613
- [Background] Shipman KL, Zeman J. Socialization of children's emotion regulation in mother-child dyads: a developmental psychopathology perspective. Dev Psychopathol. 2001 Spring;13(2):317-36. doi: 10.1017/s0954579401002073. PMID 11393649
- [Background] Nolen-Hoeksema S, Morrow J. A prospective study of depression and posttraumatic stress symptoms after a natural disaster: the 1989 Loma Prieta Earthquake. J Pers Soc Psychol. 1991 Jul;61(1):115-21. doi: 10.1037//0022-3514.61.1.115. PMID 1890582
- [Background] Weisz JR, Southam-Gerow MA, McCarty CA. Control-related beliefs and depressive symptoms in clinic-referred children and adolescents: developmental differences and model specificity. J Abnorm Psychol. 2001 Feb;110(1):97-109. doi: 10.1037//0021-843x.110.1.97. PMID 11261405
- [Background] Orpinas P, Horne AM; Multisite Violence Prevention Project. A teacher-focused approach to prevent and reduce students' aggressive behavior: the GREAT Teacher Program. Am J Prev Med. 2004 Jan;26(1 Suppl):29-38. doi: 10.1016/j.amepre.2003.09.016. PMID 14732185
- [Background] Bagby RM, Parker JD, Taylor GJ. The twenty-item Toronto Alexithymia Scale--I. Item selection and cross-validation of the factor structure. J Psychosom Res. 1994 Jan;38(1):23-32. doi: 10.1016/0022-3999(94)90005-1. PMID 8126686
- [Background] Aarons GA. Mental health provider attitudes toward adoption of evidence-based practice: the Evidence-Based Practice Attitude Scale (EBPAS). Ment Health Serv Res. 2004 Jun;6(2):61-74. doi: 10.1023/b:mhsr.0000024351.12294.65. PMID 15224451
- [Background] Weisz JR, Vaughn-Coaxum RA, Evans SC, Thomassin K, Hersh J, Ng MY, Lau N, Lee EH, Raftery-Helmer JN, Mair P. Efficient Monitoring of Treatment Response during Youth Psychotherapy: The Behavior and Feelings Survey. J Clin Child Adolesc Psychol. 2020 Nov-Dec;49(6):737-751. doi: 10.1080/15374416.2018.1547973. Epub 2019 Jan 18. PMID 30657721
- [Background] Achenbach TM. International findings with the Achenbach System of Empirically Based Assessment (ASEBA): applications to clinical services, research, and training. Child Adolesc Psychiatry Ment Health. 2019 Jul 5;13:30. doi: 10.1186/s13034-019-0291-2. eCollection 2019. PMID 31312253
- [Background] Jensen PS, Eaton Hoagwood K, Roper M, Arnold LE, Odbert C, Crowe M, Molina BS, Hechtman L, Hinshaw SP, Hoza B, Newcorn J, Swanson J, Wells K. The services for children and adolescents-parent interview: development and performance characteristics. J Am Acad Child Adolesc Psychiatry. 2004 Nov;43(11):1334-44. doi: 10.1097/01.chi.0000139557.16830.4e. PMID 15502592
- [Background] Weisz JR. Contingency and control beliefs as predictors of psychotherapy outcomes among children and adolescents. J Consult Clin Psychol. 1986 Dec;54(6):789-95. doi: 10.1037//0022-006x.54.6.789. No abstract available. PMID 3794023
- [Background] Weisz JR, Stipek DJ. Competence, contingency, and the development of perceived control. Hum Dev. 1982;25(4):250-81. doi: 10.1159/000272812. No abstract available. PMID 7141442
- [Derived] Harmon SL, Price MA, Corteselli KA, Lee EH, Metz K, Bonadio FT, Hersh J, Marchette LK, Rodriguez GM, Raftery-Helmer J, Thomassin K, Bearman SK, Jensen-Doss A, Evans SC, Weisz JR. Evaluating a Modular Approach to Therapy for Children With Anxiety, Depression, Trauma, or Conduct Problems (MATCH) in School-Based Mental Health Care: Study Protocol for a Randomized Controlled Trial. Front Psychol. 2021 Mar 5;12:639493. doi: 10.3389/fpsyg.2021.639493. eCollection 2021. PMID 33746857